CLINICAL TRIAL: NCT04490837
Title: Rapid Diagnostic Test for COVID-19 Based on Antibody Detection
Brief Title: Rapid Diagnostic Test for COVID-19 Based on Antibody Detection (YCOVID)
Acronym: YCOVID
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Juan Francisco Delgado de la Poza, Senior Medical Doctor, Corporacion Parc Tauli
Other Study IDs: 2020/587
Record Dates: First submitted 2020-05-15; First posted 2020-07-29 (Actual); Last update posted 2021-07-29 (Actual); Status verified 2021-07

CONDITIONS: Covid-19
Keywords: Antibodies; Covid-19; Rapid test; RBD
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Biospecimen Retention: Samples Without DNA — Plasma or serum
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- COVID-19 positive: Patients with clinical, radiological and/or PCR positive for COVID-19 infection
  Interventions: Diagnostic Test: ELISA and Rapid test to detect antibodies against COVID-19
- Normal: Normal human serum from blood donnors before COVID-19 pandemia
  Interventions: Diagnostic Test: ELISA and Rapid test to detect antibodies against COVID-19
- Pathological controls: Patients with other positive virological serologies
  Interventions: Diagnostic Test: ELISA and Rapid test to detect antibodies against COVID-19

INTERVENTIONS:
Diagnostic Test: ELISA and Rapid test to detect antibodies against COVID-19 — Ycovid-19 aims to be a rapid diagnostic test for SARS-CoV-2 infection, which will allow a reliable diagnosis to be made in 10 minutes, and on easy-to-use devices

SUMMARY:
Ycovid-19 aims to be a rapid diagnostic test for SARS-CoV-2 infection, which will allow a reliable diagnosis to be made in 10 minutes, and on easy-to-use devices. This test will be developed using innovative technology developed at the Parc Taulí University Hospital, which increases the immunogenicity of SARS-CoV-2 differential antigens. The increased immunogenicity of these antigens will allow to detect, with a high sensitivity and specificity, the antibodies in the serum of patients infected with SARS-CoV-2. This test will serve to confirm dubious results as well as reduce false negatives from the PCR test, which will ultimately help reduce transmission of the infection.

ELIGIBILITY:
Inclusion Criteria:

* Professional from Parc Taulí University Hospital
* Patients with clinical, radiological and/or PCR COVID-19 positive

Exclusion Criteria:

* Patients or professionals who do not sign informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with COVID-19 infection Professionals of an University Hospital
Sampling Method: Probability Sample
Enrollment: 3500 (Actual)
Dates: Start 2020-06-22 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-09-30 (Actual)

PRIMARY OUTCOMES:
IgG anti-COVID-19 | From May to July
  IgG antibodies against COVID-19 RBD
IgM anti-COVID-19 | From May to July
  IgM antibodies against COVID-19 RBD
IgA anti-COVID-19 | From May to July
  IgA antibodies against COVID-19 RBD

SECONDARY OUTCOMES:
Time of onset symptoms | From May to July
COVID-19 PCR results | From May to July
  Qualitative result to clasify patients into PCR COVID-19 positive patients and PCR COVID-19 negative patients
Radiological studies | From May to July
  The presence or abcense of the typical image of the pneumonia caused by COVID-19

CONTACTS AND LOCATIONS:
Locations (1):
- Parc Tauli University Hospital, Sabadell, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Undecided